CLINICAL TRIAL: NCT03008239
Title: Effectiveness and Safety Study of the Percutaneous Optical Fibre Glucose Sensor (FiberSense) for Home Use in Diabetic and Prediabetic Individuals
Brief Title: Effectiveness and Safety Study of the Percutaneous Optical Fibre Glucose Sensor (FiberSense)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-4.5-C-01
Record Dates: First submitted 2016-12-16; First posted 2017-01-02 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FiberSense sensor (Experimental): Type 1, Type 2 and prediabetic subjects will wear one FiberSense sensor, randomly allocated to either the upper arm (50%) or abdomen (50%) for 28 days. In addition, these subjects will wear a Dexcom sensor on the other side of the abdomen for 7 days in one of the four study weeks.
  In all 4 CAPD subjects, one FiberSense sensor will be placed in the upper arm for 28 days. No additional comparator sensor will be placed in CAPD subject.
  Interventions: Device: FiberSense sensor; Device: Dexcom Sensor

INTERVENTIONS:
Device: FiberSense sensor — The FiberSense system is a glucose-monitoring device indicated for continually recording interstitial fluid glucose levels in patients ages 18 and older with insulin dependent diabetes mellitus for the purpose of improving diabetes management.
Device: Dexcom Sensor — Dexcom is a continuous glucose monitoring (CGM) system. The display device shows the glucose readings and the trend.

SUMMARY:
This study evaluates the performance and safety of the fluorescence based fibre optic glucose sensor for home usage.24 subjects will take part in the study, including 4 pre-diabetic subjects, 8 Type I diabetic patients, 8 Type II diabetic patients and 4 diabetic patients who require continuous ambulatory peritoneal dialysis (CAPD). Type 1, Type 2 and prediabetic subjects will wear one FiberSense sensor, randomly allocated to either the upper arm (50%) or abdomen (50%) for 28 days. In addition, these subjects will wear a Dexcom sensor on the other side of the abdomen for 7 days in one of the four study weeks. In all 4 CAPD subjects, one FiberSense sensor will be placed in the upper arm for 28 days. No additional comparator sensor will be placed in CAPD subjects.

DETAILED DESCRIPTION:
The FiberSense system is a glucose-monitoring device indicated for continually recording interstitial fluid glucose levels in patients ages 18 and older with insulin dependent diabetes mellitus for the purpose of improving diabetes management. The System is intended for use by patients at home and in health care facilities.

The FiberSense system is indicated for use as an adjunctive device to complement, not replace, information obtained from standard home glucose monitoring devices.

The FiberSense system aids in the detection of episodes of hyperglycemia and hypoglycemia, facilitating both acute and long-term therapy adjustments, which may minimize these excursions.

ELIGIBILITY:
Inclusion Criteria:

* Type I or II diabetes mellitus requiring insulin in the management of glucose control for at least one year prior to enrollment or diabetes on continuous ambulatory peritoneal dialysis or prediabetic individuals with impaired fasting glucose or impaired glucose tolerance by OGTT
* Male or female age ≥ 18 years old and ≤ 70 year old.
* Women who are not pregnant, lactating or planning a pregnancy during their participation in the clinical study.
* Willingness, ability and commitment to comply with the testing, procedure and follow-up outlined in this protocol including (but not limited to) frequency of clinic visits and use of pre-specified glucose monitoring devices.
* Willingness to abstain from swimming during their participation in the measurement phase.
* In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a good study candidate.
* Written informed consent to participate in the study provided by the patient.

Exclusion Criteria:

* Poorly controlled diabetes mellitus with HbA1C >11%.
* Currently pregnant, as demonstrated by a positive pregnancy test at screening and on Day00 .
* Impaired hepatic function measured as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ three times the upper reference limit.
* Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study.
* Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff.
* Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
* Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
* Have a known allergy to medical-grade adhesives, or known hypersensitivity to any of the products used in the study.
* Known current or recent alcohol or drug abuse
* Blood donation of more than 500 ml within the last three months
* Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
* Has a MRI scan, CT scan, or diathermy scheduled during the proposed study participation.
* An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).
* Women of reproductive potential who are unwilling to adopt contraceptive measures during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | 28 days
  The primary endpoint is the proportion of FiberSense readings within ≤15% of the reference (YSI) reading for blood glucose levels >100 mg/dl, and the proportion of FiberSense readings within ≤15 mg/dl of the YSI reading for blood glucose levels ≤100 mg/dl, for paired samples taken during the in-clinic sessions.
Adverse Events reporting | 35 days

SECONDARY OUTCOMES:
Mean Relatives Differences from YSI | 28 days
Median Relatives Differences from YSI | 28 days
Mean Absolute Relative Differences from YSI | 28 days
Median Absolute Relative Differences from YSI | 28 days
Hypoglycemia detection rates | 28 days
Hyperglycemia detection rates | 28 days
Accuracy of glucose rate of change of FiberSense sensor compared to glucose rate of change of YSI | 28 days
Lag time between FiberSense readings and YSI results during induced glucose excursions | 28 days
Agreement and accuracy relative to SMBG readings (same model to be used by all subjects) | 28 days
Calibration stability | 28 days
Sensor stability | 28 days
Sensor life | 28 days
User satisfaction questionnaire score | 28 days
Blood maltose concentrations | 28 days
  Measured in CAPD subjects during the V1 in-clinic session

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, Dr., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No